CLINICAL TRIAL: NCT04724837
Title: A Phase 2b Multicentre, Randomised, Double-Blind, Active-Controlled, Parallel Group Dose-Ranging Study to Assess the Efficacy, Safety and Tolerability of Zibotentan and Dapagliflozin in Patients With Chronic Kidney Disease With Estimated Glomerular Filtration Rate (eGFR) ≥ 20 mL/Min/1.73 m^2
Brief Title: Zibotentan and Dapagliflozin for the Treatment of CKD (ZENITH-CKD Trial)
Acronym: ZENITH-CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4325C00001; 2020-004101-32 (EudraCT Number)
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Disease
Keywords: Zibotentan; Nephrology; Dapagliflozin; Sodium-glucose co-transporter 2; sodium-glucose co-transporter 2 inhibitor; Kidney diseases; Endothelin antagonist
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — ZD4054; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Zibotentan Dose A + Dapagliflozin (Experimental): Participants will receive once daily oral dose A of zibotentan and 10 mg dapagliflozin for 12 weeks.
  Interventions: Drug: Zibotentan; Drug: Dapagliflozin
- Zibotentan Dose B + Dapagliflozin (Experimental): Participants will receive once daily oral dose B of zibotentan and 10 mg dapagliflozin for 12 weeks.
  Interventions: Drug: Zibotentan; Drug: Dapagliflozin
- Placebo + Dapagliflozin (Experimental): Participants will receive once daily oral dose of dapagliflozin 10 mg and placebo for 12 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Zibotentan — Participants will receive zibotentan as per the arms they are randomized.
  Arms: Zibotentan Dose A + Dapagliflozin; Zibotentan Dose B + Dapagliflozin
Drug: Dapagliflozin — Participants will receive 10 mg dapagliflozin as per the arms they are randomized.
Drug: Placebo — Participants will receive placebo as per the arms they are randomized to.
  Arms: Placebo + Dapagliflozin

SUMMARY:
The purpose of the study is to assess efficacy, safety and tolerability of treatment with zibotentan and dapagliflozin in combination and dapagliflozin 10 mg as monotherapy in participants with chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR) ≥ 20 mL/min/1.73 m^2, and urinary albumin to creatinine ratio (UACR) ≥ 150 mg/g and ≤ 5000 mg/g.

DETAILED DESCRIPTION:
The study will be conducted in approximately 220 sites in North America, South America, Africa, Asia/Pacific, and European countries.

Participants will be randomized to 12 weeks of treatment plus 2 weeks follow-up.

After screening, eligible participants will be stratified by diabetes (diabetic kidney disease [DKD] versus non-diabetes mellitus [non-DM] CKD) and baseline eGFR (below or equal versus above 45 mL/min/1.73m^2).

A total of 495 participants will be randomised into this study, including participants randomised under the earlier study design. Four hundred and fifteen (415) participants will be randomised to have 166 participants in zibotentan Dose A/dapagliflozin 10 mg combination arm and dapagliflozin 10 mg monotherapy arm, and 83 participants in the zibotentan Dose B/dapagliflozin 10 mg combination arm.

* Zibotentan Dose A + Dapagliflozin 10 mg once daily.
* Zibotentan Dose B + Dapagliflozin 10 mg once daily.
* Placebo + Dapagliflozin 10 mg once daily

Participants who were previously randomised cannot be re-randomised.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Diagnosis of Chronic kidney disease (CKD), defined as:

  (a) eGFR chronic kidney disease epidemiology collaboration (CKD-EPI) ≥ 20 mL/min/1.73 m^2, and (b) UACR ≥ 150 and ≤ 5000 mg albumin/g creatinine, based on a single first morning void spot urine sample at screening.
* No current or prior (within 1 month of screening) medical treatment with an SGLT2i (sodium-glucose co-transporter 2 inhibitor) or any fixed dose combination with SGLT2i.
* If Angiotensin-converting enzyme inhibitors (ACEi) and/or Angiotensin receptor blockers (ARB) and/or mineralocorticoid receptor agonist are prescribed, the dose must be stable ≥ 4 weeks before screening. Participants who have been deemed unable to tolerate ACEi or ARB therapy due to allergy or complications can be enrolled.
* No current or prior treatment within 6 months prior to screening with cytotoxic therapy, immunosuppressive therapy or other immunotherapy for primary or secondary kidney disease.
* Body mass index ≤ 40 kg/m^2.
* Male or female of non-childbearing potential.
* Female participants must have a negative pregnancy test at screening, must not be lactating, and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:

  * Postmenopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone and luteinizing hormone levels in the postmenopausal range.
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.
* Male participants must be surgically sterile, abstinent, or in conjunction with a female sexual partner, using a highly effective method of contraception for the duration of the study (from the time they sign consent) and for 3 months after the last dose of investigational product to prevent any pregnancies. Male study participants must not donate or bank sperm during this same time period.
* Capable of giving signed informed consent, as described in Appendix A, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Provision of signed and dated, written ICF prior to any mandatory study-specific procedures, sampling, and analyses.
* Provision of signed and dated written Genetic informed consent prior to collection of samples (optional) for genetic analysis.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Minimal change disease, unstable rapidly progressing renal disease, and/or renal disease requiring significant immunosuppression, autosomal dominant or autosomal recessive polycystic kidney disease.
* Participants with New York Heart Association classification functional heart failure (HF) class III or IV.
* Acute coronary syndrome events within 3 months prior to screening.
* Participants with a B-type natriuretic peptide (BNP) ≥ 200 pg/mL or NT-proBNP ≥ 600 pg/mL (BNP ≥ 400 pg/mL or NT-proBNP ≥ 1200 pg/mL, respectively, if associated with atrial fibrillation) measured by local laboratory at screening (Visit 1).
* Participants with unstable HF requiring hospitalisation for optimisation of HF treatment and/or who have not been stable on HF therapy within 6 months prior to screening
* Heart failure due to cardiomyopathies that would primarily require other specific treatment: eg, cardiomyopathy due to pericardial disease, amyloidosis or other infiltrative diseases, cardiomyopathy related to congenital heart disease, primary hypertrophic cardiomyopathy, cardiomyopathy related to toxic or infective conditions (ie, chemotherapy, infective myocarditis, septic cardiomyopathy).
* High output HF (eg, due to hyperthyroidism or Paget's disease).
* Heart failure due to primary cardiac valvular disease/ dysfunction, severe functional mitral or tricuspid valve insufficiency, or planned cardiac valve repair/replacement.
* Participants with uncontrolled diabetes mellitus (HbA1c > 12%).
* Participants with Type 1 diabetes mellitus.
* Hyponatremia, defined as serum Na+ < 135 mmol/L at the time of screening (Visit 1).
* Intermittent or persistent second or third degree atrioventricular block after sinus node dysfunction, with clinically significant bradycardia or sinus pause when not treated with pacemaker.
* Prolonged QT interval (QTcF > 470 ms) on ECG at screening (Visit 1) or randomisation visit (Visit 2), known congenital long QT syndrome or history of QT prolongation associated with other medications.
* History of any life-threatening cardiac dysrhythmia (continuous or paroxysmal or uncontrolled ventricular rate in participants with atrial fibrillation or atrial flutter).
* Cardiac surgery or non-elective percutaneous coronary interventions (PCI/TAVI) (within 3 months) or open chest coronary artery bypass grafting or valvular repair/replacement (within 3 months) prior to screening or is planned to undergo any of these procedures after randomisation.
* Heart transplantation or left ventricular assist device at any time.
* Kidney or any organ transplantation.
* History or ongoing allergy/hypersensitivity, as judged by the investigator, to SGLT2i (eg, dapagliflozin, canagliflozin, empagliflozin) or drugs with a similar chemical structure to zibotentan.
* Any clinically significant disease or disorder (eg, cardiovascular, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, psychiatric, major physical impairment), which might put the participant at risk because of participation in the study, or probable alternative primary reason for participant's symptoms in judgment of investigator, including but not limited to:

  * Isolated pulmonary arterial hypertension [PAP] (defined as mean PAP ≥ 25 mmHg at rest) or right ventricular failure; in the absence of left-sided HF
  * Anaemia defined as haemoglobin (Hb) level < 100 g/L or 10 g/dL at screening (Visit 1)
  * Severe chronic obstructive pulmonary disease or other lung disease including but not limited to pulmonary fibrosis requiring chronic oxygen therapy, regular nebuliser use, or oral steroid therapy
* Stroke, transient ischemic attack, carotid surgery, or carotid angioplasty within previous 3 months prior to screening.
* Severe hepatic impairment (Child-Pugh class C Hepatic impairment), aspartate transaminase or alanine transaminase > 2x the upper limit of normal [ULN]; or total bilirubin > 2x ULN at time of screening.
* Participants with newly detected pathological laboratory values or an ongoing disease condition requiring investigation and/or initiation or adjustment of current treatment (in the opinion of the investigator).
* Positive hepatitis C antibody, or hepatitis B virus, surface antigen at screening.
* Positive human immunodeficiency virus (HIV) test.
* Participants treated with strong or moderate CYP3A4 inhibitor or inducer.
* Any condition outside the renal and CV disease area, such as but not limited to malignancy, with a life expectancy of less than 2 years based on investigator's clinical judgment.
* Confirmation of corona virus disease- 2019 (COVID-19) infection:

  * Participant has a positive test result for severe acute respiratory syndrome coronavirus 2 during screening. Participants who are not hospitalised for COVID-19 infections can be re screened 4 weeks after they have recovered.
  * Participant has been previously hospitalised with COVID-19 infection.
* Ejection fraction < 50% measured by echocardiogram at screening.
* Participation in another clinical study with an investigational product administered in the last 3 months prior to screening.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
* Previous randomisation into the present study.
* Plasma donation within 1 month of the visit at the clinic or any blood donation/blood loss > 500 mL during the 3 months prior to any visit at the clinic.
* Male participant in a sexually active relation with pregnant or breastfeeding partner.
* Participants can decline to participate in the genetic research and may still participate in the study. Exclusion from this optional genetic research may be for any of the exclusion criteria specified for the main study or any of the following:

  * Previous allogeneic bone marrow transplant.
  * Non-leukocyte depleted whole blood transfusion within 120 days of genetic sample collection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Wheeler, MB ChB, MD, FRCP, Principal Investigator — Centre for Nephrology Royal Free Campus University College London Rowland Hill Street London NW3 2PF United Kingdom; Jamie P. Dwyer, M.D., Principal Investigator — Nephrology Clinical Trials Center Nephrology and Hypertension Vanderbilt University Medical Center Nashville TN United States of America
Locations (144):
- United States (47):
  - Research Site, Huntsville, Alabama
  - Research Site, Beverly Hills, California
  - Research Site, Downey, California
  - Research Site, Fountain Valley, California
  - Research Site, Laguna Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Ontario, California
  - Research Site, South Gate, California
  - Research Site, Tarzana, California
  - Research Site, Vacaville, California
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Orlando, Florida
  - Research Site, Riverview, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Fayetteville, Georgia
  - Research Site, Wichita, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Metairie, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Flint, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Greenville, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Marion, Ohio
  - Research Site, Chester, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Conroe, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Odessa, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Waxahachie, Texas
  - Research Site, Forest, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Spokane, Washington
- Argentina (9):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Junín
  - Research Site, Mar del Plata
  - Research Site, San Luis
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Australia (5):
  - Research Site, Adelaide
  - Research Site, Birtinya
  - Research Site, Elizabeth Vale
  - Research Site, Gosford
  - Research Site, Westmead
- Brazil (7):
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (7):
  - Research Site, Gabrovo
  - Research Site, Kozloduy
  - Research Site, Montana
  - Research Site, Plovdiv
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (4):
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
- Croatia (2):
  - Research Site, Pula
  - Research Site, Vinkovci
- Denmark (3):
  - Research Site, Århus N
  - Research Site, Gentofte Municipality
  - Research Site, Roskilde
- Georgia (6):
  - Research Site, Batumi
  - Research Site, Gori
  - Research Site, Gurjaani
  - Research Site, Kutaisi
  - Research Site, Marneuli
  - Research Site, Tbilisi
- Hungary (3):
  - Research Site, Debrecen
  - Research Site, Hatvan
  - Research Site, Miskolc
- Italy (6):
  - Research Site, Bari
  - Research Site, Genova
  - Research Site, Germaneto
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, San Giovanni Rotondo
- Japan (10):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Koshigaya-shi
  - Research Site, Nagoya
  - Research Site, Naka
  - Research Site, Osaka
  - Research Site, Takarazuka-shi
  - Research Site, Tsu
  - Research Site, Ueda-shi
  - Research Site, Yakushi
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Dordrecht
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Oświęcim
  - Research Site, Poznan
  - Research Site, Rzeszów
- Research Site, Rimavská Sobota, Slovakia
- South Africa (7):
  - Research Site, Bellville
  - Research Site, Bloemfontein
  - Research Site, Durban
  - Research Site, George
  - Research Site, Observatory
  - Research Site, Pretoria
  - Research Site, Somerset West
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Burela de Cabo
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Seville
  - Research Site, Valencia
- Ukraine (9):
  - Research Site, Chernivtsі
  - Research Site, Dnipro
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhia
  - Research Site, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Smeijer JD, Wasehuus VS, Dhaun N, Gorriz JL, Soler MJ, Astrand M, Mercier AK, Greasley PJ, Ambery P, Heerspink HJL. Effects of Zibotentan Alone and in Combination with Dapagliflozin on Fluid Retention in Patients with CKD. J Am Soc Nephrol. 2024 Oct 1;35(10):1381-1390. doi: 10.1681/ASN.0000000000000436. Epub 2024 Jul 12. PMID 39352861
- [Derived] Heerspink HJL, Kiyosue A, Wheeler DC, Lin M, Wijkmark E, Carlson G, Mercier AK, Astrand M, Ueckert S, Greasley PJ, Ambery P. Zibotentan in combination with dapagliflozin compared with dapagliflozin in patients with chronic kidney disease (ZENITH-CKD): a multicentre, randomised, active-controlled, phase 2b, clinical trial. Lancet. 2023 Nov 25;402(10416):2004-2017. doi: 10.1016/S0140-6736(23)02230-4. Epub 2023 Nov 3. PMID 37931629
- [Derived] Heerspink HJL, Greasley PJ, Ahlstrom C, Althage M, Dwyer JP, Law G, Wijkmark E, Lin M, Mercier AK, Sunnaker M, Turton M, Wheeler DC, Ambery P. Efficacy and safety of zibotentan and dapagliflozin in patients with chronic kidney disease: study design and baseline characteristics of the ZENITH-CKD trial. Nephrol Dial Transplant. 2024 Feb 28;39(3):414-425. doi: 10.1093/ndt/gfad183. PMID 37632201
- [Derived] Smeijer JD, Kohan DE, Webb DJ, Dhaun N, Heerspink HJL. Endothelin receptor antagonists for the treatment of diabetic and nondiabetic chronic kidney disease. Curr Opin Nephrol Hypertens. 2021 Jul 1;30(4):456-465. doi: 10.1097/MNH.0000000000000716. PMID 33990507
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4325C00001&attachmentIdentifier=76401f22-ca7c-4db3-afd7-6421e415f203&fileName=redacted_Protocol.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4325C00001&attachmentIdentifier=d582702a-ca97-4d99-8960-313ecc5880b0&fileName=redacted_SAP.pdf&versionIdentifier=
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4325C00001&attachmentIdentifier=15320161-ea3a-4aee-b08c-65187b046cd1&fileName=redacted_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in approximately 170 sites in North America, South America, Africa, Asia/Pacific, and European countries.
Pre-assignment Details: The screening period was of 4 weeks. All the study assessments were performed as per the schedule of assessments. Participants who met the eligibility criteria were randomised to study intervention. The reason of discrepancy between enrollment number versus subjects in the full analysis set and safety analysis set is that not all randomized subjects were included in analysis. Enrollment number is 542 when number of subjects included in the full analysis set and safety analysis set is 447.
Groups:
- Zibotentan 0.25 mg + Dapagliflozin: Participants received once daily oral dose of 0.25 mg zibotentan and 10 mg dapagliflozin for 12 weeks.
- Zibotentan 1.5 mg + Dapagliflozin: Participants received once daily oral dose of 1.5 mg zibotentan and 10 mg dapagliflozin for 12 weeks.
- Placebo + Dapagliflozin: Participants received once daily oral dose of dapagliflozin 10 mg and matching placebo for 12 weeks.
Period: Overall Study
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
Started | 91 | 179 | 177
Full Analysis Set | 91 | 179 | 177
Safety Analysis Set | 91 | 179 | 177
Completed | 82 | 142 | 157
Not Completed | 9 | 37 | 20
Not completed — Other | 4 | 16 | 0
Not completed — Withdrawal by Subject | 2 | 9 | 9
Not completed — Adverse Event | 2 | 7 | 4
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Failure to Meet Randomization Criteria | 0 | 1 | 3
Not completed — Study Terminated by Sponsor | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who were randomised and received any study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin | Total
Number analyzed (Participants) | 91 | 179 | 177 | 447
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (12.72) | 62.7 (12.33) | 63.6 (11.60) | 62.8 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 55 | 55 | 138
  Male | 63 | 124 | 122 | 309
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 58 | 46 | 127
  Not Hispanic or Latino | 68 | 121 | 131 | 320
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 18 | 26 | 26 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 7 | 17 | 22 | 46
  White | 56 | 124 | 125 | 305
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Albumin to Creatinine Ratio (UACR) From Baseline to Week 12
Description: The effect of zibotentan 1.5/dapagliflozin 10 mg versus dapagliflozin 10 mg on UACR was assessed.
Time Frame: From baseline (Week 0 [Day 1]) until Week 12 (Day 84)
Population: The full analysis set included all participants who were randomised and received any study intervention. Here, N = number of participants analyzed refers to n = number analyzed for this outcome measure at specific timepoints.
Measure: Geometric Mean (Standard Error); unit: milligram/gram (mg/g)
Arm/Group | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
Number analyzed (Participants) | 105 | 132
milligram/gram (mg/g) | 0.48 (1.094) | 0.72 (1.090)
Statistical Analysis 1: Comparison: Zibotentan 1.5 mg + Dapagliflozin vs Placebo + Dapagliflozin; Comparison between Zibotentan 1.5 mg + Dapagliflozin and Dapagliflozin 10 mg + Placebo (PBO); Test type: Superiority — Two-sided p-value is presented. A p-value <0.10 indicates statistical significance, which is consistent with a one-sided test at the 5% level; p < 0.001, Mixed Models Analysis; Adjusted % mean change from baseline = -33.7, 90% CI 2-sided [-42.5 to -23.5] — If adjusted percentage mean change from baseline >0 then the result favours Dapa 10 mg + PBO for UACR

2. Secondary Outcome: Change in UACR From Baseline to Week 12
Description: The effect of zibotentan 0.25 mg/dapagliflozin 10 mg versus dapagliflozin 10 mg monotherapy on UACR was assessed.
Time Frame: From baseline (Week 0 [Day 1]) until Week 12
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: mg/g
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Placebo + Dapagliflozin
Number analyzed (Participants) | 62 | 132
mg/g | 0.52 (1.106) | 0.72 (1.090)
Statistical Analysis 1: Comparison: Zibotentan 0.25 mg + Dapagliflozin vs Placebo + Dapagliflozin; Comparison between Zibotentan 0.25 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.002, Mixed Models Analysis; Adjusted % mean change from baseline = -27.0, 90% CI 2-sided [-38.4 to -13.6] — If adjusted percentage mean change from baseline >0 then the result favours Dapa 10 mg + PBO for UACR

3. Secondary Outcome: Change in Office Systolic Blood Pressure From Baseline to Week 12
Description: The change in office systolic blood pressure for doses of zibotentan combined with dapagliflozin 10 mg versus dapagliflozin 10 mg monotherapy was assessed.
Time Frame: From baseline (Week 0 [Day 1]) until Week 12 (Day 84)
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Millimeters of mercury (mmHg)
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
Number analyzed (Participants) | 65 | 108 | 137
Millimeters of mercury (mmHg) | -7.1 [-10.0 to -4.1] | -11.0 [-13.5 to -8.4] | -3.4 [-5.8 to -1.0]
Statistical Analysis 1: Comparison: Zibotentan 0.25 mg + Dapagliflozin vs Placebo + Dapagliflozin; Comparison between Zibotentan 0.25 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; Least Square (LS) mean CFB = -3.6, 90% CI 2-sided [-6.8 to -0.5] — If mean change from baseline (CFB) >0 then the result favours Dapa 10 mg + PBO for office systolic blood pressure
Statistical Analysis 2: Comparison: Zibotentan 1.5 mg + Dapagliflozin vs Placebo + Dapagliflozin; Comparison between Zibotentan 1.5 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean CFB = -7.6, 90% CI 2-sided [-10.3 to -4.9] — If mean change from baseline >0 then the result favours Dapa 10 mg + PBO for office systolic blood pressure

4. Secondary Outcome: Change in Office Diastolic Blood Pressure From Baseline to Week 12
Description: The change in office diastolic blood pressure for doses of zibotentan combined with dapagliflozin 10 mg versus dapagliflozin 10 mg monotherapy was assessed.
Time Frame: From baseline (Week 0 [Day 1]) until Week 12 (Day 84)
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: mmHg
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
Number analyzed (Participants) | 65 | 108 | 137
mmHg | -4.3 [-6.2 to -2.5] | -6.8 [-8.4 to -5.2] | -1.4 [-2.9 to 0.1]
Statistical Analysis 1: Comparison: Zibotentan 0.25 mg + Dapagliflozin vs Placebo + Dapagliflozin; Comparison between Zibotentan 0.25 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS Mean CFB = -3.0, 90% CI 2-sided [-5.0 to -1.0] — If mean change from baseline >0 then the result favours Dapa 10 mg + PBO for office diastolic blood pressure
Statistical Analysis 2: Comparison: Zibotentan 1.5 mg + Dapagliflozin vs Placebo + Dapagliflozin; Comparison between Zibotentan 1.5 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS Mean CFB = -5.4, 90% CI 2-sided [-7.1 to -3.7] — If mean change from baseline >0 then the result favours Dapa 10 mg + PBO for office diastolic blood pressure

5. Secondary Outcome: Change in UACR From Baseline to Week 12
Description: The assessment of dose-response and relationship across different dose of zibotentan/dapagliflozin and dapagliflozin alone on UACR reduction.
Time Frame: From baseline (Week 0 [Day 1]) until Week 12 (Day 84)
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: mg/g
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
Number analyzed (Participants) | 62 | 105 | 132
mg/g | 0.52 (1.106) | 0.48 (1.094) | 0.72 (1.090)
Statistical Analysis 1: Comparison: Zibotentan 0.25 mg + Dapagliflozin vs Placebo + Dapagliflozin; Comparison between Zibotentan 0.25 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; Adjusted % mean change from baseline = -27.0, 90% CI 2-sided [-38.4 to -13.6] — If adjusted percentage mean change from baseline >0 then the result favours Dapa 10 mg + PBO for UACR
Statistical Analysis 2: Comparison: Zibotentan 1.5 mg + Dapagliflozin vs Placebo + Dapagliflozin; Comparison between Zibotentan 1.5 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; Adjusted % mean change from baseline = -33.7, 90% CI 2-sided [-42.5 to -23.5] — If adjusted percentage mean change from baseline >0 then the result favours Dapa 10 mg + PBO for UACR

6. Secondary Outcome: Change in eGFR From Baseline to Week 1, Week 12, and Week 14
Description: The effect of different doses of zibotentan and dapagliflozin 10 mg in combination versus dapagliflozin 10 mg monotherapy on eGFR was assessed.
Time Frame: From baseline (Week 0 [Day 1]) until Week 1 (Day 8), Week 12 (Day 84), and Week 14 (Day 98)
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: milliliters/minutes/1.73 square metres
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
Number analyzed (Participants) | 83 | 152 | 151
milliliters/minutes/1.73 square metres
  Week 1 | -2.0 [-3.5 to -0.5] | -3.9 [-5.2 to -2.6] | -3.1 [-4.4 to -1.8]
  Week 12: number analyzed (Participants) | 64 | 108 | 135
  Week 12 | -3.1 [-4.7 to -1.5] | -3.0 [-4.4 to -1.6] | -1.9 [-3.3 to -0.6]
  Week 14: number analyzed (Participants) | 63 | 105 | 131
  Week 14 | 0.2 [-1.4 to 1.8] | -2.0 [-3.4 to -0.6] | 0.1 [-1.2 to 1.5]
Statistical Analysis 1: Comparison: Zibotentan 0.25 mg + Dapagliflozin vs Placebo + Dapagliflozin; Week 1 - Comparison between Zibotentan 0.25 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean CFB = 1.1, 90% CI 2-sided [-0.5 to 2.6] — If mean change from baseline <0 then the result favours Dapa 10 mg + PBO for eGFR
Statistical Analysis 2: Comparison: Zibotentan 1.5 mg + Dapagliflozin vs Placebo + Dapagliflozin; Week 1 - Comparison between Zibotentan 1.5 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean CFB = -0.8, 90% CI 2-sided [-2.1 to 0.5] — If mean change from baseline <0 then the result favours Dapa 10 mg + PBO for eGFR
Statistical Analysis 3: Comparison: Zibotentan 0.25 mg + Dapagliflozin vs Placebo + Dapagliflozin; Week 12 - Comparison between Zibotentan 0.25 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean CFB = -1.2, 90% CI 2-sided [-2.8 to 0.5] — If mean change from baseline <0 then the result favours Dapa 10 mg + PBO for eGFR
Statistical Analysis 4: Comparison: Zibotentan 1.5 mg + Dapagliflozin vs Placebo + Dapagliflozin; Week 12 - Comparison between Zibotentan 1.5 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean CFB = -1.1, 90% CI 2-sided [-2.5 to 0.3] — If mean change from baseline <0 then the result favours Dapa 10 mg + PBO for eGFR
Statistical Analysis 5: Comparison: Zibotentan 0.25 mg + Dapagliflozin vs Placebo + Dapagliflozin; Week 14 - Comparison between Zibotentan 0.25 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean CFB = 0.1, 90% CI 2-sided [-1.6 to 1.8] — If mean change from baseline <0 then the result favours Dapa 10 mg + PBO for eGFR
Statistical Analysis 6: Comparison: Zibotentan 1.5 mg + Dapagliflozin vs Placebo + Dapagliflozin; Week 14 - Comparison between Zibotentan 1.5 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean CFB = -2.1, 90% CI 2-sided [-3.5 to -0.7] — If mean change from baseline <0 then the result favours Dapa 10 mg + PBO for eGFR

7. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: The safety and tolerability of all doses of zibotentan combined with dapagliflozin 10 mg and dapagliflozin 10 mg monotherapy was assessed.
Time Frame: From Screening (Day -28) until Follow-up visit (Day 98), up to 126 days
Population: The safety analysis set included all participants that were randomised and received any study intervention. Here, N = number of participants analyzed refers to n = number analyzed for this outcome measure at specific timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
Number analyzed (Participants) | 91 | 179 | 177
Participants
  Any AE | 45 | 86 | 66
  AE with outcome of death | 0 | 0 | 1
  Any SAE | 2 | 10 | 4
  Any AE leading to discontinuation of investigational product (IP) | 11 | 22 | 7
  Any AE leading to dose interruption | 3 | 7 | 10
  Any AE leading to withdrawal from study | 2 | 7 | 4
  Any AE possibly related to IP | 14 | 33 | 16

8. Secondary Outcome: Change in eGFR From Week 1 to Week 12
Description: as for outcome 6
Time Frame: From Week 1 (Day 8) to Week 12 (Day 84)
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: milliliters/minutes/1.73 square metres
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
Number analyzed (Participants) | 64 | 108 | 135
milliliters/minutes/1.73 square metres | -1.1 [-2.5 to 0.4] | 0.9 [-0.2 to 2.0] | 1.2 [0.1 to 2.2]
Statistical Analysis 1: Comparison: Zibotentan 0.25 mg + Dapagliflozin vs Placebo + Dapagliflozin; Week 1 and Week 12 - Comparison between Zibotentan 0.25 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean change = -2.2, 90% CI 2-sided [-4.0 to -0.4] — If mean change <0 then the result favours Dapa 10 mg + PBO for eGFR
Statistical Analysis 2: Comparison: Zibotentan 1.5 mg + Dapagliflozin vs Placebo + Dapagliflozin; Week 1 and 12 - Comparison between Zibotentan 1.5 mg + Dapagliflozin and Dapagliflozin 10 mg + PBO; Test type: Superiority; Mixed Models Analysis; LS mean change = -0.3, 90% CI 2-sided [-1.8 to 1.3] — If mean change <0 then the result favours Dapa 10 mg + PBO for eGFR

ADVERSE EVENTS:
Time Frame: From screening (Day -28) to Final Follow-up (Day 98), up to 126 days
Arm/Group | Zibotentan 0.25 mg + Dapagliflozin | Zibotentan 1.5 mg + Dapagliflozin | Placebo + Dapagliflozin
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/179 | 1/177
Serious Adverse Events (participants affected / at risk) | 2/91 | 10/179 | 4/177
Other Adverse Events (participants affected / at risk) | 14/91 | 24/179 | 6/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zibotentan 0.25 mg + Dapagliflozin (N=91) | Zibotentan 1.5 mg + Dapagliflozin (N=179) | Placebo + Dapagliflozin (N=177)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zibotentan 0.25 mg + Dapagliflozin (N=91) | Zibotentan 1.5 mg + Dapagliflozin (N=179) | Placebo + Dapagliflozin (N=177)
Metabolic acidosis (Metabolism and nutrition disorders) | 5 (5) | 7 (8) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 8 (9) | 2 (2)
Hypertension (Vascular disorders) | 5 (5) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 2 (2) | 9 (9) | 1 (1)

LIMITATIONS AND CAVEATS:
No multiple testing correction was considered in this early phase study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT04724837/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT04724837/SAP_003.pdf